CLINICAL TRIAL: NCT04122430
Title: Risk of Venous Thromboembolism in Patients Receiving First-Line Chemotherapy for Disseminated Germ Cell Tumours - a Multi-Site Retrospective Cohort Study as Part of the Global Germ-Cell Cancer Group (G3) Consortium
Brief Title: Risk of Venous Thromboembolism in Patients Receiving First-Line Chemotherapy for Disseminated Germ Cell Tumours
Acronym: G3 RPLN PBC
Status: Completed | Type: Observational
Sponsor: Walter and Eliza Hall Institute of Medical Research (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other); Melbourne Health (Other)
Responsible Party: Principal Investigator, Dr Ben Tran, Medical Oncologist/Clinical Researcher, Walter and Eliza Hall Institute of Medical Research
Other Study IDs: QA2015168
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Testicular Neoplasms
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- GCT treated with first line chemotherapy: Men with disseminated Germ Cell Tumours-GCT (AJCC Stage IS, 2, or 3) and have received first line chemotherapy with curative intent for disseminated GCT
  .
  Interventions: Other: Review of Health Information

INTERVENTIONS:
Other: Review of Health Information

SUMMARY:
Recent data (Srikanthan and Tran et al. JCO 2014, in press) have demonstrated that the presence of large retroperitoneal lymph node metastases on baseline staging scans (measuring >5cm in axial dimension) are associated with significantly increased risk of venous thromboembolism in patients receiving first line chemotherapy for disseminated germ cell tumours.

This study, a G3 collaborative effort, aims to confirm these findings in a large multi-national validation cohort.

DETAILED DESCRIPTION:
Recent data (Srikanthan and Tran et al. JCO 2014, in press) have demonstrated that the presence of large retroperitoneal lymph node (RPLN) metastases on baseline staging scans (measuring >5cm in axial dimension) are associated with significantly increased risk of venous thromboembolism (VTE) in patients receiving first line chemotherapy for disseminated germ cell tumours (GCT).

This study, a G3 collaborative effort, aims to confirm these findings in a large multi-national validation cohort.

Primary objective:

To validate the association between large RPLN metastases (measuring >5cm in axial dimension) and increased risk of VTE during and immediately after completion of (within 90 days) first line chemotherapy for disseminated GCT.

Secondary objectives:

* To assess the discriminatory accuracy for VTE of both large RPLN metastases and high-risk Khorana score (defined as > 3)
* To determine the incidence of VTE in patients with disseminated GCT receiving first line chemotherapy at baseline, during chemotherapy and immediately following chemotherapy
* To determine the incidence of VTE during and immediately after chemotherapy in patients receiving prophylactic anticoagulation during first line chemotherapy for disseminated GCT
* To determine the incidence of major bleeding in patients who received prophylactic anticoagulation versus those who did not
* To determine overall survival at 12 months, 3 years and 5 years for patients who developed VTE compared to those who did not No identifying data (e.g. name, hospital UR, address) will be collected.

Data will be collected by retrospective review of the medical chart.

When assessing for the presence of large RPLN as a risk factor for VTE, only the maximal diameter of the long axis of the largest retroperitoneal lymph node metastasis will be recorded. Where the exact measurement is not available, it should be recorded whether the maximal diameter of the largest RPLN measures >5cm or <5cm. The representative value for large RPLN should NOT include the combination of all maximal diameters of all RPLN metastases.

Regarding the pre-chemotherapy values for hemoglobin, platelet count and leukocyte count, these must have been conducted within 30 days of initiation of chemotherapy. The highest serum Creatinine observed during the course of chemotherapy should also be recorded - this is not necessarily the pre-chemotherapy serum Creatinine, as the highest value may have occurred during chemotherapy.

A VTE event is defined as either deep vein thrombosis (DVT) or pulmonary embolism (PE). Superficial venous thrombosis or thrombophlebitis will not be considered as a VTE event. Only bleeding events requiring medical intervention will be recorded.

Data collection will cover the period from the start of curative first line chemotherapy until 90 days following completion of chemotherapy. Any VTE event that is present at baseline (i.e. start of first line chemotherapy) will be recorded. Additionally, any VTE event that occurs within 90 days of completion of chemotherapy will be recorded; this allows recording of incidental VTE noted on post-chemotherapy restaging scans. Distinction will be made for VTE that occurs following post-chemo surgery (post-op) that is performed within the 90 day timeframe.

Data collection should be completed by December 31, 2015 and de-identified data forwarded to the Principal Investigator for data analysis before January 30, 2015.

The aggregated data will be used for study reports, and where appropriate conference presentations and peer-reviewed manuscript(s). In addition, the findings may be used to inform the design of a subsequent prospective trial of prophylactic anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

1. Men with disseminated GCT (AJCC Stage IS, 2, or 3)
2. Received first line chemotherapy with curative intent for disseminated GCT
3. Clinical data available from chemotherapy initiation to at least 90 days following completion of chemotherapy (patients who died prior to 90 days will be included in this study)
4. Initiated chemotherapy between 1-January-2000 and 31-December-2014* *Data collection from consecutive patients initiating chemotherapy during a defined period within the specified timeframe is acceptable (e.g. patient data from 5-year period starting 1-January-2008 and ending 31-December-2012 is acceptable)

Exclusion Criteria:

1. Prior chemotherapy for GCT (including use of adjuvant chemotherapy or curative chemotherapy for prior diagnosis of disseminated GCT).
2. History of secondary malignancy (excluding non-melanoma superficial skin cancers)

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Men with disseminated GCT (AJCC Stage IS, 2, or 3) who have received first line chemotherapy with curative intent for disseminated GCT.
  Clinical data available from chemotherapy initiation to at least 90 days following completion of chemotherapy (patients who died prior to 90 days will be included in this study) and initiated chemotherapy between 1-January-2000 and 31-December-2014.
Sampling Method: Non-Probability Sample
Enrollment: 1135 (Actual)
Dates: Start 2015-12; Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
To validate the association between large RPLN metastases (measuring >5cm in axial dimension) and increased risk of VTE during and immediately after completion of (within 90 days) first line chemotherapy for disseminated GCT | March 2016

SECONDARY OUTCOMES:
To assess the discriminatory accuracy for VTE of both large RPLN metastases and high-risk Khorana score (defined as > 3) | March 2016
To determine the incidence of VTE in patients with disseminated GCT receiving first line chemotherapy at baseline, during chemotherapy and immediately following chemotherapy | March 2016
To determine the incidence of VTE during and immediately after chemotherapy in patients receiving prophylactic anticoagulation during first line chemotherapy for disseminated GCT | March 2016
To determine the incidence of major bleeding in patients who received prophylactic anticoagulation versus those who did not | March 2016
To determine overall survival at 12 months, 3 years and 5 years for patients who developed VTE compared to those who did not. | March 2016

CONTACTS AND LOCATIONS:
Overall Officials: Ben Tran, Medicine, Principal Investigator — Walter and Eliza Hall Institute of Medical Resaerch
Locations (1):
- Walter and Eliza Hall Institute of Medical Research, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No